CLINICAL TRIAL: NCT01725048
Title: A Pilot Study to Evaluate Individualized Choice of Antidepressant in Patients With Cancer
Brief Title: Pilot Study to Evaluate Individualized Choice of Antidepressants in Patients With Cancer
Acronym: NRR
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: LCCC 1021
Record Dates: First submitted 2012-11-07; First posted 2012-11-12 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Major Depressive Disorder; Neoplasms
Keywords: Major depressive disorder; Neoplasms
MeSH Terms: conditions — Depressive Disorder, Major; Neoplasms | interventions — Mirtazapine; Citalopram

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mirtazapine (Active Comparator): Treatment with oral mirtazapine, dosed once daily, for 9 weeks, with starting dose of 7.5 milligrams (mg) daily up to 30mg daily.
  Interventions: Drug: Mirtazapine
- Citalopram (Active Comparator): Treatment with Citalopram, once daily, for 9 weeks, with dosages starting at 10mg once daily to 40mg once daily.
  Interventions: Drug: Citalopram

INTERVENTIONS:
Drug: Mirtazapine — 7.5mg by mouth once a day at night. If subject has not had a 50% or greater reduction in the PHQ-9 depression assessment score, and if the subject is not experiencing unacceptable adverse effects, then the dose may be escalated first to 15mg by mouth every night and then to 30mg by mouth every night.
  Other Names: Remeron
  Arms: Mirtazapine
Drug: Citalopram — Citalopram 10mg by mouth once daily. If the subject has not had a 50% or greater reduction in PHQ-9 depression assessment score, and if the subject is not experiencing unacceptable side effects, then the dose may be escalated first to 20mg by mouth every day and then to 40mg by mouth once a day.
  Other Names: Celexa
  Arms: Citalopram

SUMMARY:
This is a pilot study to test the hypothesis that the antidepressants mirtazapine and citalopram are effective treatment for major depressive disorder (MDD) in cancer patients.

DETAILED DESCRIPTION:
Major depressive disorder (MDD) is a debilitating illness associated with increased mortality and significant impairment in quality of life. The prevalence of MDD is particularly high in patients with cancer, as much as 38% in some studies.

The study of depression in cancer patients is particularly important, as these co-morbid illnesses can frequently complicate the management of each other. In addition to affecting quality of life, poorly controlled depression can affect cancer treatment adherence and can lead to poor treatment outcomes.

Depression can be challenging to diagnose in patients with cancer. A spectrum of depressive symptoms can be seen, ranging from appropriate sadness in response to a life threatening diagnosis, to a major depressive episode. The diagnosis is confounded by the symptoms brought on by the cancer and its treatment, such as fatigue, insomnia, anorexia, and pain. Medications commonly used in cancer patients such as narcotics, benzodiazepines, antihistamines, steroids, antibiotics, chemotherapy, and endocrine therapy can all lead to side effects that further confuse the picture. However, while challenging, evidence does suggest that a valid diagnosis of depression can be made in this patient population.

The current standard for diagnosing MDD is the Diagnostic and Statistical Manual of Mental Disorders - Fourth Edition - Text Revision (DSM-IV-TR), which was published in 2000 by the American Psychiatric Association. The diagnosis is made based on an interview between the patient and physician in which nine criteria are assessed, including depressed mood, anhedonia, weight loss or gain, insomnia or hypersomnia, psychomotor agitation or retardation, fatigue, feelings of worthlessness or guilt, difficulty concentrating, and recurrent thoughts of death. In patients with cancer, the diagnosis of MDD is more often based on anhedonia and feelings of worthlessness, as depressed mood, weight fluctuation, and sleep disturbance can be symptoms of the underlying cancer itself. Once the diagnosis has been made, there are several tools which have been created and validated for the purpose of assessing the severity of depression and for following the severity over time. The tool we intend to use in this study is the PHQ-9.

Therapy for MDD in the general population includes both psychotherapy and pharmacological intervention. However, the optimal therapy of MDD in cancer patients remains uncertain. Very few placebo controlled trials have been performed in this population, and there is currently no uniformly accepted standard of care. Some of the evidence from studies in depressed but otherwise medically healthy patients may be applicable to cancer patients, but there are several factors which complicate the treatment of depression in this group. For example, the overlap of symptoms between depression and the underlying malignancy can confound the diagnosis, as discussed earlier. Simultaneous treatment of the underlying malignancy introduces adverse effects from surgery, chemotherapy, or radiation, as well as an increased likelihood of drug-drug interactions. Finally, co-morbid conditions such as cancer pain can contribute to the depression, requiring simultaneous therapy. As a result of these unique factors, the treatment of MDD in cancer patients cannot necessarily be approached using the standard recommendations for the general population.

There is scant evidence supporting the effectiveness of pharmacologic therapy in cancer patients with MDD. In the last 25 years only four placebo controlled trials have been published, and of these only two have shown a statistically significant improvement in depression scores with active treatment.

Additional studies are needed to evaluate some of the newer antidepressants within the cancer population and to assess whether this strategy of matching side effects to symptoms is beneficial.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with a malignancy
* Informed consent obtained and signed
* Greater than or equal to 18 years of age
* Life expectancy determined to be greater than or equal to 6 months
* Diagnosed with Major Depressive Disorder based on clinical examination and the DSM-IV-TR criteria
* PHQ-9 depression assessment completed by subject, with a score of 10 or greater
* Able to take whole or crushed tablets by mouth or by feeding tube

Exclusion Criteria:

* Unable to complete self-report instruments due to illiteracy, neurologic illness, visual problems, inability to speak or read English, or other causes
* Treatment with antidepressants or antipsychotics within the last 3 months
* Psychotic or manic behavior
* Active suicidal ideation or plan
* Current illicit substance abuse
* Severe renal impairment as defined by creatinine clearance of <15 milliliters/minute/1.73 meters squared (mL/min/m2)
* Severe hepatic impairment as defined by Aspartate Aminotransferase (AST) or alanine aminotransferase (ALT) >5x the upper limit of normal, or a total bilirubin > 3.0 milliliters/deciliter (mL/dL)
* History of congenital long QT syndrome
* Clinically significant congestive heart failure or bradyarrhythmias
* Treatment with a concomitant medication that is known to have a strong association with corrected QT interval (QTc) prolongation AND a QTc >460 for men or >470 for women. Applicable to the citalopram arm only

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-01; Primary Completion 2012-05 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Feasibility | One year
  To determine the feasibility of this pilot study to recruit subjects, as measured by the number of individuals enrolled per month, such that the goal of the study is met in a timely manner.

SECONDARY OUTCOMES:
Depression Score | 9 weeks
  To assess the short-term (9 week) outcome of mirtazapine or citalopram in cancer patients with major depressive disorder based on mean improvement in depressive symptoms as measured by the Patient Health Questionnaire (PHQ-9)

CONTACTS AND LOCATIONS:
Overall Officials: Eliza Park, MD, Principal Investigator — University of North Carolina
Locations (1):
- University of North Carolina Hospital, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Vita G, Compri B, Matcham F, Barbui C, Ostuzzi G. Antidepressants for the treatment of depression in people with cancer. Cochrane Database Syst Rev. 2023 Mar 31;3(3):CD011006. doi: 10.1002/14651858.CD011006.pub4. PMID 36999619
- See also: Website for the University of North Carolina Lineberger Comprehensive Cancer Center — http://www.unclineberger.org
- See also: Website for the National Cancer Institute — http://www.cancer.gov